CLINICAL TRIAL: NCT05761886
Title: Rural Area Pharmacist Intervention for Diabetes - Management Using eHealth: A Pilot Study (RAPID-ME)
Brief Title: Rural Area Pharmacist Intervention for Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00094019
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes
Keywords: Telehealth; Rural populations; Clinical pharmacy services
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: the target sample size in our pilot study is 72 in the intervention group. The target for the control group is 168.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telehealth-based clinical pharmacy intervention (Experimental): will involve a pharmacist identifying and addressing medication-related problems (e.g., inappropriate dosage or indications, drug interactions, and therapeutic duplication); optimizing medication regimens (discontinuing if appropriate, providing subsidized and generic options, and reducing medication complexity); and providing T2D education and self-management support
  Interventions: Other: telehealth-based clinical pharmacy intervention
- usual care (No Intervention): will involve routine physician office visits every 3 (for those with HbA1c outside goal) - or every 6 months (for those with HbA1c within goal). Medication regimens are usually managed by physicians, nurse practitioners, and physician assistants, and Patients have access to centralized chronic disease management programs.

INTERVENTIONS:
Other: telehealth-based clinical pharmacy intervention — The pharmacist will perform an initial comprehensive review of the medication regimen, make any adjustments, document those in the patient's electronic health record (EHR) and communicate with the patient's T2D care team as needed. They will also call (using an EHR-based software) the patient using phone/video to educate them about T2D self-management and identify any medication-related unmet needs. Periodic reviews of the medication regimen and roughly biweekly follow-up patient calls will occur with frequency based on need (as judged by the pharmacist). Patient intervention calls will be personalized depending on HbA1c levels, comorbidities, and medication complexity
  Arms: telehealth-based clinical pharmacy intervention

SUMMARY:
The goal of the project is to inform the system leaders regarding the feasibility and utility of having an embedded telehealth-based clinical pharmacist at rural primary care practices for supportive disease management of patients with Type 2 diabetes (T2D) and whether continuing and expanding the program within the system is worthwhile.

DETAILED DESCRIPTION:
Improvement of suboptimal type 2 diabetes (T2D) management and outcomes in rural areas in the United States (US) is an urgent national health policy priority. Novel approaches such as telehealth and supportive clinical management of T2D by non-physician providers have been recommended to fill gaps in care. With specialty in drug therapy, clinical pharmacists are in a position to uniquely contribute to filling gaps in T2D management related to medication therapy, which are common and often the cause of adverse outcomes in patients with T2D. The objective of this pilot study is to determine the feasibility, acceptability, appropriateness, fidelity, barriers and facilitators of implementation, and preliminary effectiveness of a telehealth-based clinical pharmacy intervention to inform the design of a subsequently planned fully powered effectiveness-implementation trial of the intervention. This pilot study will involve randomization based on the days the patients had encounters at participating practices (4 in North Carolina). The 2 study arms will be: 1) Usual care, receiving standard practice of care managed by physicians, nurse practitioners, and physician assistants with access to chronic disease management services and 2) Intervention arm, receiving the intervention consisting of clinical pharmacy services including identification and resolution of medication-related problems and patient needs, optimization of medication regimen and T2D education and self-management support, in addition to usual care. The intervention will last for 3 months and will consist of biweekly video/phone calls between patients and the pharmacist. Based on recommendations from literature on pilot studies, the total planned sample size is 240 patients. Implementation science framework by Proctor and colleagues and scales by Weiner and colleagues (for feasibility, acceptability, appropriateness, and fidelity) and Consolidated Framework for implementation Research (for barriers and facilitators of intervention implementation) will guide collection of data on outcomes. for using complementary medicine and healthcare avoidance. The results of our work will facilitate wide implementation of the intervention and thereby improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years and <=75 years (since children have different incidence, management, and outcomes of Type 2 diabetes (T2D) compared to adults and older adults aged more than 75 years may have had their hemoglobin A1C (HbA1c) goals adjusted to higher thresholds)
* HbA1c reading ≥ 8% recorded during 6 months prior to or up to 9 days after the encounter at the participating practices
* Uncontrolled type 2 diabetes (ICD-10-CM code E11.XX) recorded in the EHR in the year prior to up to 1 week after the uncontrolled HbA1c reading

Exclusion Criteria:

* Patients with gestational or type 1 diabetes
* Those enrolled in any other chronic disease management programs delivered by non-physician healthcare professionals
* Those receiving T2D care from an endocrinologist
* Those receiving long term, hospice, or palliative care services
* Those with serious mental illnesses (schizophrenia and other psychotic disorders, major depressive disorders, bipolar disorders, and borderline personality disorder)
* Those with malignant cancer
* Those with cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Patient enrollment rates | Month 13
  Proportion of eligible patients enrolled
Proportion of patients with complete data | Month 17
  Proportion of patients with complete data
Proportion of respondents selecting a response - Feasibility | Month 17
  Proportion of respondents selecting a response of agree/strongly agree (disagree/strongly disagree for negatively worded items) on 70% of the survey items measuring perspectives regarding whether it was possible for the respondents to perform the program activities
Proportion of respondents selecting a response - Acceptability | Month 17
  Proportion of respondents selecting a response of agree/strongly agree (disagree/strongly disagree for negatively worded items) on 70% of the survey items measuring perspectives regarding whether they approve and like the program
Proportion of respondents selecting a response - Appropriateness | Month 17
  Proportion of respondents selecting a response of agree/strongly agree (disagree/strongly disagree for negatively worded items) on 70% of the survey items measuring perspectives regarding program fit with the needs of the respondents
Proportion of items self-reported by pharmacist - Fidelity | Month 17
  Proportion of items self-reported by pharmacist by checking (yes/no/not applicable) in a task-list of program activities

SECONDARY OUTCOMES:
Change in HbA1c | Month 17
  Change in HbA1c from baseline to follow-up - While the usually recommended HbA1c target is <7.0%, the American Diabetes Association recommends transitioning the HbA1c target to ≥8.0% based on factors such as age, limited life expectancy, complications, history of hypoglycemia, and comorbidities.
Change in Blood Pressure | Month 17
  Change in systolic and diastolic blood pressure from baseline to follow-up - A normal blood pressure can vary between individuals, but the American Heart Association recommend a target blood pressure below 120 mm Hg systolic and 80 mm Hg diastolic. Usually, hypertension is defined as blood pressure above 140/90 and is considered severe if the pressure is above 180/120.
Number of Acute Care Days | Month 17
  Change in the number of days spent in emergency room or hospital from baseline to follow-up
Change in patient-reported medication adherence scores | Month 17
  Change in patient-reported medication adherence score from baseline to follow-up measured by a survey
  Change in patient-reported medication adherence score from baseline to follow-up measured by a single item survey: "Over the past week, what percent of the time did you take all your diabetes medications as your doctor prescribed?" [11 response categories (0, 10, 20... 100%) with higher score indicating better adherence]
Change in barriers to medication adherence | Month 17
  Change in patient-reported barriers to medication adherence score from baseline to follow-up
  Adherence Starts with Knowledge-12 survey - measured by Adherence Starts with Knowledge-12 survey (Score can range from 12-60, with higher scores representing greater barriers to adherence.)

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Mahabaleshwarkar, PhD, Principal Investigator — Atrium Health Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-02-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT05761886/ICF_000.pdf